CLINICAL TRIAL: NCT07370155
Title: A Phase 1, Open-Label, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Migaldendranib (MGB) in Healthy Volunteers
Brief Title: Study Evaluating Safety & Tolerability of Migaldendranib in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ashvattha Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D-4517-003
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Myoglobin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MGB 200 mg (Experimental): Participants receive MGB 200 mg administered subcutaneously once weekly on Days 1, 8, and 15 to evaluate safety, tolerability, and pharmacokinetics.
  Interventions: Drug: MGB 200 mg
- MGB 400 mg (Experimental): Participants receive MGB 400 mg administered subcutaneously once weekly on Days 1, 8, and 15 following Safety Review Committee approval.
  Interventions: Drug: MGB 400 mg
- MGB 600 mg (Experimental): Participants receive MGB 600 mg administered subcutaneously once weekly on Days 1, 8, and 15, contingent upon acceptable safety and tolerability in prior cohorts.
  Interventions: Drug: MGB 600 mg

INTERVENTIONS:
Drug: MGB 200 mg — Participants receive weekly subcutaneous administration of MGB
  Arms: MGB 200 mg
Drug: MGB 400 mg — Participants receive an intermediate dose of MGB administered subcutaneously once weekly
  Arms: MGB 400 mg
Drug: MGB 600 mg — Participants receive the highest planned dose of MGB administered subcutaneously
  Arms: MGB 600 mg

SUMMARY:
This is a Phase 1, open-label, multiple-dose study to evaluate the safety, tolerability, and PK of MGB after weekly subQ MGB administration in up to 36 healthy volunteers at 1 site in Australia.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multiple-dose study to evaluate the safety, tolerability, and pharmacokinetics (PK) of MGB administered following weekly subcutaneous dosing in healthy adult volunteers. Up to 36 participants will be enrolled at a single site in Australia.

The study includes a screening period of up to 27 days, an 18-day treatment period, and follow-up visits on Days 22 and 29. Participants will be enrolled into up to six sequential dose-escalation cohorts (up to six participants per cohort) using a sentinel dosing approach. Dosing includes weekly subcutaneous administration of MGB at escalating doses.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy man or woman age 18 to 65 years, inclusive, at the Screening Visit
2. Has the ability to understand and sign the written ICF and local medical privacy authorization forms, which must be obtained prior to any study-related procedures being completed
3. Is in general good health, based upon the results of a medical history assessment, physical examination, vital signs, and laboratory profile, as judged by the Investigator
4. Female participants of non-childbearing potential must be either surgically sterile (hysterectomy, bilateral tubal ligation, salpingectomy, and/or bilateral oophorectomy at least 26 weeks before the Screening Visit) or postmenopausal, defined as spontaneous amenorrhea for at least 1 year, with follicle-stimulating hormone (FSH) in the postmenopausal range at screening, based on the central laboratory's ranges
5. All female participants of childbearing potential with male partners and male participants with female partners of childbearing potential must consent to use 2 (two) highly effective methods of contraception from start of study and for at least 90 days following the EOS visit or last dose of study treatment, whichever is later. Women of childbearing potential on hormonal contraceptives must be stable on the medication for at least 2 menstrual cycles prior to Day -1.

   The following are acceptable methods of highly effective contraception:
   * Using twice the normal protection of birth control by using a condom AND one other form of contraception; either birth control pills (The Pill), or injectable birth control, birth control patch or contraceptive implant associated with inhibition of ovulation, or intrauterine device; or
   * Surgical sterilization as a single form of birth control: i.e., tubal ligation, hysterectomy, bilateral oophorectomy, vasectomy, or equivalently effective surgical form of birth control (with documented proof of the absence of sperm in the post-vasectomy ejaculate) at least 6 months prior to screening; or
   * True sexual abstinence for the duration of the study and for at least 12 weeks following the EOS visit or after the last dose of IP, whichever is later, is acceptable only when in line with the preferred and usual lifestyle of the participant.
   * Periodic abstinence (calendar, symptothermal, post ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea methods are not considered "true" abstinence and are not acceptable methods of contraception.
6. If male, participants must agree to abstain from sperm donation through 90 days after administration of the last dose of study drug
7. If female, participants must refrain from donation of ova from start of study and for 120 days after last dose of investigational drug
8. Female participants may not be pregnant, lactating, or breastfeeding
9. Female participants of childbearing potential must have a negative pregnancy test at screening and Check-in (Day -1)
10. Participants must have a negative test result for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVab), and human immunodeficiency virus (HIV) antibody at screening
11. Participants must have an estimated glomerular filtration rate (eGFR) of 90 mL/min/1.73 m2 at screening
12. Participants must have a negative urine test for drugs of abuse (see Appendix B), cotinine, and breath alcohol test at screening and Check-in (Day -1)
13. Participants must be willing and able to abide by all study requirements and restrictions.

Exclusion Criteria:

1. Evidence of clinically significant hematologic, renal, endocrine, pulmonary, cardiac, gastrointestinal (GI), hepatic, psychiatric, neurologic, immunologic, allergic disease (including multiple or clinically significant drug allergies), or any other condition that, in the opinion of the Investigator, might significantly interfere with the absorption, distribution, metabolism, or excretion of study drug, or place the participant at an unacceptable risk as a participant in this study
2. Evidence of systemic inflammation as measured by C-reactive protein above the upper limit of normal, as measured by the local lab
3. History of malignancy (other than successfully treated basal cell or squamous cell skin cancer)
4. History or presence of an abnormal electrocardiogram (ECG) that, in the opinion of the Investigator, is clinically significant
5. Laboratory results (serum chemistry, hematology, coagulation, and urinalysis) outside the normal range at screening and Check-in and considered clinically significant in the opinion of the Investigator. Any elevation of aspartate transaminase (AST) and alanine transaminase (ALT) above the upper limit of normal at screening and/or Check-in is exclusionary. One retest of an exclusionary laboratory result is allowed at the discretion of the Investigator
6. Has had an acute illness considered clinically significant by the Investigator within 30 days prior to screening
7. History of alcoholism or drug abuse within 1 year prior to screening or excessive alcohol consumption defined as >14 standard drinks per week.
8. Has used any product containing nicotine within 30 days prior to screening or intends to use any product containing nicotine during the study (exception of ≤ 5 cigarettes per week)
9. Has had any immunizations (live vaccines) in the 4 weeks prior to screening; COVID-19 vaccination within 7 days of Day 1
10. Has used any prescription (with the exception of hormonal contraceptives) or over-the counter medication (with the exception of acetaminophen), vitamins/herbal supplements within7 days prior to Day 1
11. Has used any other study drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to Day 112. Has lost or donated > 450 mL of whole blood or blood products within 7 days prior to screening

13. Investigator has reason to believe that the participant may be unable to fulfill the protocol visit schedule or requirements 14. Has any finding that, in the view of the Investigator or Medical Monitor, would compromise the participant's safety requirements 15. Is employed by the Sponsor, the Contract Research Organization (CRO), or the study site (permanent, temporary contract worker, or designee responsible for the conduct of the study), or is a family member (spouse, parent, sibling, or child) of the Sponsor, CRO, or study site employee

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-29 (Estimated); Primary Completion 2026-05-13 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of MGB | Varying timepoints through end of treatment, up to approximately 22 days.
  Safety will be assessed throughout the study by monitoring adverse events (AEs), including their incidence, severity, and relationship to study treatment. Additional safety assessments will include clinical laboratory evaluations (hematology, clinical chemistry, and urinalysis), physical examinations, and vital sign measurements, including pulse rate, blood pressure (BP), respiration rate, and tympanic temperature.

SECONDARY OUTCOMES:
Pharmacokinetic Parameter Area Under the Curve (AUC) for MGB | Varying timepoints through end of treatment, up to approximately 22 days.
  Measure of MGB AUC in plasma
Pharmacokinetic Parameter Maximum Concentration (Cmax) for MGB | Varying timepoints through end of treatment, up to approximately 22 days.
  Measure of MGB Cmax in plasma
Pharmacokinetic Parameter Time to Maximum Concentration (Tmax) for MGB | Varying timepoints through end of treatment, up to approximately 22 days.
  Measure of MGB Tmax in plasma
Pharmacokinetic Parameter Total Clearance (CL) for MGB | Varying timepoints through end of treatment, up to approximately 22 days.
  Measure of MGB CL in plasma
Pharmacokinetic Parameter Apparent Terminal Half-life (t1/2) for MGB | Varying timepoints through end of treatment, up to approximately 22 days.
  Measure of MGB Apparent Terminal Half-life (t1/2) in plasma

IPD SHARING:
Plan to Share IPD: No